CLINICAL TRIAL: NCT03442036
Title: A Randomized, Observer-Masked, Controlled, Parallel-Arm, Clinical Trial Comparing Through-the-Needle With Suture-Method Perineural Catheter Designs for Continuous Popliteal-Sciatic Nerve Blocks
Brief Title: Comparing Through-the-Needle With Suture-Method Catheter Designs for Popliteal Nerve Blocks
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: Ferrosan Medical Devices, Roskilde, Denmark (Industry)
Responsible Party: Principal Investigator, Brian M. Ilfeld, MD, MS, Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Suture vs Standard Catheters
Record Dates: First submitted 2018-02-15; First posted 2018-02-22 (Actual); Results first posted 2020-03-12 (Actual); Last update posted 2021-02-17 (Actual); Status verified 2021-01

CONDITIONS: Regional Anesthesia; Sciatic Nerve Block
Keywords: Regional Anesthesia; Sciatic Nerve Block; Continuous Nerve Block; Perineural Catheter

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized using a computer-generated list and opaque, sealed envelopes to one of two treatment groups (blocks of 4, no stratification): perineural catheter insert using (1) through-the-needle technique or (2) suture technique.
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Through-the-Needle Technique (Active Comparator): Perineural catheters are inserted through a straight hollow-bore needle.
  The perineural catheter will then be used to infuse local anesthetic directly onto the nerve to provide postoperative pain control.
  Interventions: Device: Through-the-Needle Technique
- Suture-Method Technique (Experimental): Perineural catheters are attached to the back of a hollow suture-shaped needle that pulls the catheter adjacent to the target nerve.
  The perineural catheter will then be used to infuse local anesthetic directly onto the nerve to provide postoperative pain control.
  Interventions: Device: Suture-Method Technique

INTERVENTIONS:
Device: Suture-Method Technique — Perineural catheters are attached to the back of a hollow suture-shaped needle that pulls the catheter adjacent to the target nerve
  Arms: Suture-Method Technique
Device: Through-the-Needle Technique — Perineural catheters are inserted through a straight hollow-bore needle
  Arms: Through-the-Needle Technique

SUMMARY:
Following painful surgical procedures, postoperative analgesia is often provided with a single-injection peripheral nerve block. Hothe investigatorsver, even with the longest-acting FDA-approved local anesthetic currently available-bupivacaine-the block duration is measured in hours, while the surgical pain may persist for days. A continuous peripheral nerve block allows a prolonged block, consisting of a percutaneously-inserted catheter with its orifice adjacent to a target nerve/plexus through which local anesthetic may be administered. Two basic perineural catheter designs currently exist: (1) catheters that are inserted either through or over a straight hollow-bore needle; and, (2) catheters that are attached to the back of a hollow suture-shaped needle that pulls the catheter adjacent to the target nerve ("suture-method" design). To date, a comparison of the relative risks and benefits of these two designs have not been investigated. The investigators therefore propose a randomized, observer-masked, controlled, parallel-arm, clinical trial to compare these two catheter designs when used to provide post-surgical analgesia following foot and ankle surgery.

DETAILED DESCRIPTION:
This investigation will be a randomized, observer-masked, controlled, parallel-arm, human-subjects clinical trial. Of note, the investigators will be using standard-of-care perineural catheters and local anesthetic under their FDA-approved purpose and do not plan to research a possible change of indication or use of these drugs as part of this research project.

Consenting adults undergoing surgery with a planned popliteal-sciatic perineural catheter placement will be offered enrollment. Study inclusion will be proposed to eligible patients prior to surgery. If a patient desires study participation, written, informed consent will be obtained using a current UCSD IRB-approved ICF.

Following written, informed consent, the investigators will collect baseline anthropomorphic information (age, sex, height, and the investigatorsight). Subjects will be then be randomized using a computer-generated list and opaque, sealed envelopes to one of two treatment groups (blocks of 4, no stratification): perineural catheter insertion using (1) through-the-needle technique or (2) suture technique. All catheters will be placed by a regional anesthesia fellow or resident under the direct supervision and guidance of a regional anesthesia attending (or by the attending him/herself).

All subjects will have a peripheral intravenous (IV) catheter inserted, standard noninvasive monitors applied, supplemental oxygen administered via a nasal cannula or face mask, and positioned prone. Midazolam and fentanyl (IV) will be titrated for patient comfort, while ensuring that patients remain responsive to verbal cues. The area that will be subsequently covered by the catheter dressing will be clipped of hair, if necessary. The ultrasound will be placed to visualize the short axis (cross-section) of the sciatic nerve to identify the sciatic nerve bifurcation which will subsequently be marked, as well as the location 5 cm cephalad to the bifurcation. The area will be cleaned with chlorhexidine gluconate and isopropyl alcohol and a clear, sterile, fenestrated drape applied. The ultrasound probe will be placed to visualize the short-axis (cross-section) of the target nerve(s) and the target for the catheter to intercept the nerve may be anywhere between the bifurcation and 5 cm cephalad to the bifurcation. All catheters will be placed using standard UCSD ultrasound-guided perineural catheter techniques as previously described. Normal saline 5-20 mL will be administered via the needle and/or catheter to allow catheter insertion and/or testing of catheter location (viewed with ultrasound).

Local anesthetic (20 mL, lidocaine 2% with epinephrine 1:200,000-400,000) will be administered via the catheter. A "successful" catheter insertion will be defined as sensory-block onset in the tibial nerve distribution within 30 minutes following the local anesthetic injection. If the nerve block fails, the catheter will be replaced or the patient removed from further study.

An infusion pump will be attached to the patient's perineural catheter and initiated within the recovery room. The pump will provide ropivacaine 0.2% at a 6 mL/h basal rate infusion and a 4 mL patient-controlled bolus with a 30 minute lockout (standard at UCSD). Subjects will be discharged with a prescription for oxycodone 5 mg tablets for supplementary analgesia. Subjects will be contacted via phone for 4 days following surgery to collect study outcome measures: worst, average, least, and current surgical pain (Numeric Rating Scale of 0 to 10, with "0" being no pain and "10" being the worst pain ever experienced), analgesic use (oral opioids and infusion boluses), sleep disturbances, opioid and local anesthetic infusion side effects, local anesthetic leakage, gross catheter dislodgement, sensory and motor block, and satisfaction with pain control. Subjects or their caretakers will remove the catheters at home.

Primary endpoint:

Hypothesis 1: Surgical pain will be noninferior within the first 2 days following foot/ankle surgery with a suture-method compared with a through-the-needle perineural catheter when used for a continuous popliteal-sciatic nerve block to provide postoperative analgesia (the mean "average" pain measured daily with a Numeric Rating Scale).

Hypothesis 2: Opioid consumption will be noninferior within the first 2 days following foot/ankle surgery with a suture-method compared with a through-the-needle perineural catheter when used for a continuous popliteal-sciatic nerve block to provide postoperative analgesia (cumulative dose).

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing ambulatory foot or ankle surgery with a popliteal perineural catheter for postoperative analgesia.

Exclusion Criteria:

* Pregnancy
* Inability to communicate with research staff
* Incarceration
* Clinically apparent neuropathy in the operative extremity
* Chronic high dose opioid use
* History of opioid abuse
* Concurrent surgery outside the block distribution
* Patients with nerves deeper than 5 cm from the skin

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2018-04-06 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-04-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John J Finneran IV, MD, Study Director — UC San Diego; Brian M Ilfeld, MD, MS, Principal Investigator — UC San Diego
Locations (1):
- UCSD Medical Center, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects undergoing painful foot/ankle surgery at UCSD were recruited to the study. Total enrollment = 70 subjects.
Groups:
- Through-the-Needle Technique: Perineural catheters were inserted through a straight hollow-bore needle.
  The perineural catheter was then used to infuse local anesthetic directly onto the nerve to provide postoperative pain control.
- Suture-Method Technique: Perineural catheters are attached to the back of a hollow suture-shaped needle that pulls the catheter adjacent to the target nerve.
  The perineural catheter was then used to infuse local anesthetic directly onto the nerve to provide postoperative pain control.
Period: Overall Study
Arm/Group | Through-the-Needle Technique | Suture-Method Technique
Started | 35 | 35
Completed | 35 | 35
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Through-the-Needle Technique: Perineural catheters are inserted through a straight hollow-bore needle.
  The perineural catheter will then be used to infuse local anesthetic directly onto the nerve to provide postoperative pain control.
  Through-the-Needle Technique: Perineural catheters are inserted through a straight hollow-bore needle
- Suture-Method Technique: Perineural catheters are attached to the back of a hollow suture-shaped needle that pulls the catheter adjacent to the target nerve.
  The perineural catheter will then be used to infuse local anesthetic directly onto the nerve to provide postoperative pain control.
  Suture-Method Technique: Perineural catheters are attached to the back of a hollow suture-shaped needle that pulls the catheter adjacent to the target nerve
- Total: Total of all reporting groups
Arm/Group | Through-the-Needle Technique | Suture-Method Technique | Total
Number analyzed (Participants) | 35 | 35 | 70
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 35 | 26 | 61
  >=65 years | 0 | 9 | 9
Age, Continuous [Mean (Standard Deviation); unit: Years] | 37.5 (12.6) | 52.6 (16.8) | 45 (16.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 14 | 28
  Male | 21 | 21 | 42
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 35 | 35 | 70

OUTCOME MEASURES:

1. Primary Outcome: Average Pain
Description: Pain evaluated using a numeric rating scale with 0 = no pain and 10 = worst imaginable pain
Time Frame: first two postoperative days combined
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Through-the-Needle Technique | Suture-Method Technique
Number analyzed (Participants) | 35 | 35
score on a scale | 2.7 (2.4) | 3.4 (2.4)

2. Secondary Outcome: Opioid Consumption
Description: Cumulative opioid consumption (oxycodone) measured in milligrams
Time Frame: first two postoperative days
Measure: Median (Inter-Quartile Range); unit: milligrams
Arm/Group | Through-the-Needle Technique | Suture-Method Technique
Number analyzed (Participants) | 35 | 35
milligrams
  Postoperative Day 1 | 5.0 [0 to 15] | 10 [0 to 20]
  Postoperative Day 2 | 10 [0 to 20] | 10 [0 to 20]

3. Secondary Outcome: Worst Pain
Description: The worst pain score for the day evaluated using a numeric rating scale with 0 = no pain and 10 = worst imaginable pain
Time Frame: Postoperative Days 1 and 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Through-the-Needle Technique | Suture-Method Technique
Number analyzed (Participants) | 35 | 35
score on a scale
  Postoperative Day 1 | 5.4 (3.8) | 5.8 (3.4)
  Postoperative Day 2 | 5.6 (2.9) | 5.6 (3.1)

4. Other Pre Specified Outcome: Catheter Dislodgment.
Description: We will also test for noninferiority of the suture method to the through-the-needle perineural catheter on gross catheter dislodgment using a 1-tailed noninferiority test.
Time Frame: first two postoperative days
Measure: Count of Participants; unit: Participants
Arm/Group | Through-the-Needle Technique | Suture-Method Technique
Number analyzed (Participants) | 35 | 35
Participants | 3 | 0

ADVERSE EVENTS:
Time Frame: 1 year
Groups:
- Through-the-Needle Technique: 19 Gauge Perineural catheter inserted via a 17 Gauge Touhy Neede
- Suture-Catheter: 19 Gauge Perineural catheter via 19 G Suture needle
Arm/Group | Through-the-Needle Technique | Suture-Catheter
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/35 | 1/35
Other Adverse Events (participants affected / at risk) | 0/35 | 0/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Through-the-Needle Technique (N=35) | Suture-Catheter (N=35)
Deep vein thrombosis (Vascular disorders) | 0 | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-22): https://cdn.clinicaltrials.gov/large-docs/36/NCT03442036/Prot_SAP_000.pdf